CLINICAL TRIAL: NCT05205356
Title: VIGOR: Virtual Genome Center for Infant Health
Status: Recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Boston Medical Center (Other); Baystate Medical Center (Other); UMass Memorial Health (Other); The Cooper Health System (Other); National Human Genome Research Institute (NHGRI) (NIH); DHR Health Institute for Research and Development (Other); The Hospitals of Providence East Campus (Unknown); The Hospitals of Providence Memorial Campus (Unknown); Jackson Health System (Other); University of Texas (Other); Driscoll Children's Hospital (Other); University of South Alabama (Other)
Responsible Party: Principal Investigator, Timothy Yu, Associate Professor of Pediatrics, Boston Children's Hospital
Other Study IDs: IRB-P00040496; 1R01HG011798-01A1 (NIH)
Record Dates: First submitted 2022-01-05; First posted 2022-01-25 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Genetics Disease; Genetics/Birth Defects; Genetic Predisposition to Disease
Keywords: Genetics
MeSH Terms: conditions — Genetic Diseases, Inborn; Congenital Abnormalities; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Genomic sequencing of neonates and biological parents will be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neonates and Parents/Caregivers: Providers caring for newborns that meet eligibility criteria will approach parents to assess interest. The VIGOR study staff will remotely contact parents to complete consent for genomic sequencing (GS). We will also invite 1 additional primary caregiver (e.g. father, co-mother etc.) to participate even if that caregiver is not biologically related to the child.
  We will administer surveys at baseline enrollment to assess sociodemographics, obstetrical history, family genetic history & mental health; within 1 week of disclosure of findings to assess satisfaction & mental health; & at 3 & 6 months to further assess mental health & newborn clinical outcomes. We will approach a subset of the families for qualitative interviews to assess satisfaction with VIGOR & receipt of GS results with their physician in more detail.
- Clinicians: Following focus groups at each of the participating sites to assess the feasibility & needs of each site, the care teams will receive basic training in genomics and how to disclose GS results with VIGOR support. Study orientation will be completed as part of the training. Focus groups will be conducted within 1 year post implementation & again between year 4 & the completion of the study, to assess feasibility & appropriateness of VIGOR. We will administer brief surveys to the care providers before & after receipt of genomic education to assess their baseline knowledge & comfort with genomic medicine in newborns. Surveys will be repeated within a week of disclosure to families regarding feedback on the process & satisfaction with VIGOR. After approximately 3-5 disclosure events, study staff will approach the clinical care team members to participate in a qualitative interview to assess their perspectives in more depth.

SUMMARY:
This study will provide rigorous evaluation of implementing a virtual genome center into community clinical settings without highly specialized resources, thereby offering generalizable insights as to how best to implement genomic medicine at scale and for other age groups. This intervention has great potential to address disparities in genomic medicine among low-income and underrepresented minority (URM) populations and will enhance capacity for providers and health systems to utilize highly specialized genomic techniques in their communities.

The goal of this study is to achieve equitable access to state-of-the-art genomic medical care to sick newborns in community centers that predominately care for low-income and racial/ethnic minority populations through the creation of a virtual genome center (VIGOR). VIGOR will provide a venue for physician and family education, genomic expert consultation, reanalysis of unsolved sequencing data, and access to cutting edge therapeutic innovation, thereby facilitating institutionalization of genomic best practices in community settings, and not just highly specialized referral centers.

DETAILED DESCRIPTION:
Genomic medicine has rapidly advanced in the past decade enabling earlier diagnosis and personalized treatment. However, only a few highly specialized centers in the US have the resources to take advantage of these advances in patient care. This has created a large health equity gap whereby patients cared for in typical community settings, often low-income and/or representing racial/ethnic minorities, do not receive equitable medical care. Another barrier to the wider utilization of genomic medicine is the poor dissemination of knowledge among clinicians, especially in community settings. A wide gap exists in the implementation of genomic medicine from diagnosis to personalized therapies, a field experiencing huge advances but still subject to wide disparities in accessibility. This study aims to develop and test the implementation of a strategy to break down these barriers to genomic medicine. The target population is sick newborns admitted to the NICU that present with probable genetic conditions. This study proposes a novel center, VIrtual GenOme CenteR (VIGOR). VIGOR will be a center that can remotely support clinicians and families working in community NICUs.

This study will provide rigorous evaluation of implementing a virtual genome center at community clinical settings without highly specialized resources, thereby offering generalizable insights as to how best to implement genomic medicine at scale and for other age groups. This intervention has great potential to address disparities in genomic medicine among low-income and underrepresented minorities (URM) populations and will enhance capacity for providers and health systems to utilize highly specialized genomic techniques in their communities.

The goal of this study is to achieve equitable access to state-of-the-art genomic medical care to sick newborns in community centers that predominately care for low-income and racial/ethnic minority populations through the creation of a virtual genome center (VIGOR). VIGOR will provide a venue for physician and family education, genomic expert consultation, reanalysis of unsolved sequencing data, and access to cutting edge therapeutic innovation, thereby facilitating institutionalization of genomic best practices in community settings, and not just highly specialized referral centers.

ELIGIBILITY:
Inclusion Criteria:

* Newborns presenting with probable genetic conditions inpatient on the NICU. These may include (but is not limited to) those with unexplained hypotonia, seizures, metabolic disorders, disorders of sex development, interstitial lung disease, immunodeficiency or multiple congenital anomalies.
* Babies must have at least one biologic parent available for consent and participation.
* The criteria for inclusion are 100% phenotype based and do not include any demographic parameters.

Exclusion Criteria:

* Presence of a likely nongenetic explanation for the phenotype (e.g., perinatal asphyxia explained by uterine rupture or placental pathology;
* Clinical features pathognomonic for a recognizable chromosomal abnormality, such as trisomy 21;
* Associations already known to have low genetic diagnostic yield, including VATER/VACTERL association and OEIS complex;
* Infants who die before enrollment;
* Known family history of genetic disease that is plausibly the cause of the infant's illness; - Those with a prenatal genetic diagnosis.

Ages: 0 Days to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The VIGOR center will enroll and follow for 12 months 250 eligible newborns and their families within community NICUs in the US serving diverse populations. Among enrolled newborns, rapid genomic sequencing will be facilitated along with the creation and return of timely Clinical Interpretive Reports to families and providers. This study comprehensively examine implementation outcomes according to a well-established framework at the NICU, provider, and newborn/caregiver-level.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2022-03-22 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Implementation of VIGOR | 4 year
  Penetration of VIGOR measured by percentage of eligible participants who were enrolled, tested, providers received CIR and completed a disclosure session.

SECONDARY OUTCOMES:
Implementation of VIGOR | 4 year
  Appropriateness of VIGOR measured at the provider level by conducting focus groups/interviews.
Implementation of VIGOR | 4 year
  Feasibility of VIGOR measured at the provider level by conducting focus groups/interviews.
Service Outcomes | 4 years
  Equity in penetration of VIGOR use by race/ethnicity, insurance status and primary language measured at the participant level by conducting chart reviews and surveys.
Client Outcomes | 4 years
  Function measured at the infant/caregiver and provider level by conducting surveys, chart reviews and focus groups/interviews.
Client Outcomes | 4 years
  Symptomatology measured at the infant/caregiver level by conducting surveys, and interviews.
Client Outcomes | 4 years
  Satisfaction measured at the infant/caregiver and provider level by conducting surveys, chart reviews and focus groups/interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Yu, MD, PhD, Principal Investigator — Boston Children's Hospital
Locations (10):
- United States (10):
  - USA Children's and Women's Hospital, Mobile, Alabama
  - Holtz Children's Hospital at Jackson Memorial Medical Center, Miami, Florida
  - Boston Medical Center, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - UMass Memorial Hospital, Worcester, Massachusetts
  - Cooper University Hospital, Camden, New Jersey
  - Driscoll Children's Hospital Rio Grande Valley, Edinburg, Texas
  - The Women's Hospital at Renaissance, Edinburg, Texas
  - The Hospitals of Providence, El Paso, Texas
  - University of Texas Medical Branch, Galveston, Texas

REFERENCES:
- [Derived] D'Gama AM, Hills S, Douglas J, Young V, Genetti CA, Wojcik MH, Feldman HA, Yu TW, G Parker M, Agrawal PB; VIGOR Network. Implementation of rapid genomic sequencing in safety-net neonatal intensive care units: protocol for the VIrtual GenOme CenteR (VIGOR) proof-of-concept study. BMJ Open. 2024 Feb 6;14(2):e080529. doi: 10.1136/bmjopen-2023-080529. PMID 38320840